CLINICAL TRIAL: NCT01485900
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Hemodynamics of Ascending Repeated Oral Doses of SAR407899A in Patients With Moderate Chronic Kidney Disease on Stable Angiotensin Converting Enzyme-inhibitor (ACE-I) Treatment
Brief Title: Repeated Dosing Study to Assess Safety and Tolerability in CKD-3 Patients on Stable ACE-I Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDR12446; 2011-003793-83 (EudraCT Number); U1111-1123-5699 (Other: UTN)
Record Dates: First submitted 2011-11-24; First posted 2011-12-06 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Dose 1: 20 days 3-step uptitration with doses A, B, and C of SAR407899 vs. placebo
  Interventions: Drug: SAR407899A
- Cohort 2 (Experimental): Dose 2: 20 days 3-step uptitration with doses B, C and D of SAR407899 vs. placebo
  Interventions: Drug: SAR407899A

INTERVENTIONS:
Drug: SAR407899A — Pharmaceutical form:capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

* To assess the tolerability and safety of repeated oral ascending doses of SAR407899A in patients with moderate chronic kidney disease (CKD) on stable angiotensin converting enzyme-inhibitor (ACE-I)

Secondary Objectives:

* To assess in patients with moderate CKD the effect of concomitant multiple dose of SAR407899A and ACE-Is on office and 24-hr ambulatory blood pressure and heart rate
* The effect of repeated multiple doses of SAR407899A on the pharmacodynamic response to ACE-Is (AcSDKP)
* The pharmacokinetic profile of repeated oral administration of SAR407899A during co-administration of ACE-Is

DETAILED DESCRIPTION:
The total duration for this study will be around 8 weeks.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients aged between 18 and 79
* Patients with chronic kidney disease (CKD-3)
* Patients should be on stable ACE-I treatment (same type and regimen) for at least 2 months prior to screening
* Body weight between 50.0 kg and 115.0 kg inclusive if male, between 40.0 kg and 100 kg inclusive if female
* If female, patients must be permanently sterilized for more than 3 months or postmenopausal
* Having given written informed consent prior to the study.

Exclusion criteria:

* Women of child bearing potential.
* Uncontrolled clinically relevant cardiovascular, pulmonary, gastro-intestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female) or infectious disease, or signs of acute illness
* Active hepatitis, hepatic insufficiency
* Acute renal failure
* Patients requiring dialysis during the study
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician.
* Any history of orthostatic dysregulation (including but not limited to neurocardiogenic syncope, postural orthostatic tachycardia syndrome)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting Adverse Events (AEs) | 8 weeks

SECONDARY OUTCOMES:
Clinical safety laboratory measurement including hematology and biochemistry | 8 weeks
urine and blood renal function markers | 8 weeks
ECG, vital signs measurements (Heart rate and systolic and diastolic blood pressure) | 8 weeks
AcSDKP (tetrapeptide of the composition N-Acetyl-Ser-Asp-Lys-Pro) | 8 weeks
AUC | 8 weeks
Cmax | 8 weeks
t1/2z | 8 weeks
24-hr ambulatory blood pressure | Day-1, Day 14 and Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Investigational Site Number 498002, Chisinau, Moldova
- Investigational Site Number 642001, Bucharest, Romania